CLINICAL TRIAL: NCT06185361
Title: Selective Serotonin Reuptake Inhibitors, Fluoxetine Versus the Standard Oral Desmopressin for Management of Mono-symptomatic Nocturnal Enuresis. A Randomised Controlled Trial
Brief Title: Selective Serotonin Reuptake Inhibitors, Fluoxetine Versus the Standard Oral Desmopressin for Management of Mono-symptomatic Nocturnal Enuresis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdel Azim El Helaly, Assistant Professor, Fayoum University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Nocturnal Enuresis
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Nocturnal Enuresis; Enuresis; Enuresis, Nocturnal
MeSH Terms: conditions — Nocturnal Enuresis; Enuresis | interventions — Fluoxetine; Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fluoxetine (Active Comparator): selective serotonin reuptake inhibitors fluoxetine 20 mg for 12 weeks
  Interventions: Drug: Fluoxetine 20 MG
- desmopressin (Active Comparator): 0.2 mg desmopressin tablet for 12 weeks
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Fluoxetine 20 MG — fluoxetine
  Arms: fluoxetine
Drug: Desmopressin — desmopressin
  Arms: desmopressin

SUMMARY:
To determine whether there is a role for the selective serotonin reuptake inhibitors fluoxetine versus desmopressin in the treatment of nocturnal enuresis in children who have not responded to standard nonpharmacological urotherapy, and whether there are side effects involved.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 7 years
2. Severe enuresis with at least (50%) seven wet nights out of 14
3. Failed treatment
4. The enuresis alarm was either ineffective or considered impractical due to the family circumstances.

Exclusion Criteria:

1. Underlying renal, urologic, neurologic, endocrinologic, or cardiac conditions
2. Patients with psychiatric disorders and behavioral disorders including depression, attention-deficit/hyperactivity disorder.
3. Untreated constipation
4. Contraindications to fluoxetine or desmopressin treatment

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The children will be non-responders, partial responders, or full responders to therapy | three months
  The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society "ICCS definitions" (i.e., if the reduction of enuresis frequency was below or above 50% or 90%, respectively)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided